CLINICAL TRIAL: NCT07076823
Title: Safety and Efficacy of Canagliflozin in Patients With Metastatic High Microsatellite Instability (MSI-H) Colorectal Cancer: a Phase I Trial
Brief Title: Safety and Efficacy of Canagliflozin in Patients With Metastatic High Microsatellite Instability (MSI-H) Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xuelei Ma MD, Deputy Director (Medical) of the Department of Biotherapy, Cancer Center, West China Hospital, Sichuan University; Associate Director of the Stem Cell Research and Translational Research Laboratory; PhD Supervisor; Professor/Researcher, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Approval No. 729 (2025)
Record Dates: First submitted 2025-06-23; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; SGLT-2 Inhibitor
Keywords: colorectal cancer; SGLT-2 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): PD-1 Inhibitor: Tislelizumab will be administered intravenously at the recommended dose of 200 mg every 3 weeks until disease progression or intolerable toxicity occurs.
  Canagliflozin: According to the drug's prescribing information, the recommended starting dose is 100 mg once daily (qd), taken orally before the first meal of the day. For patients who tolerate 100 mg qd and have an estimated glomerular filtration rate (eGFR) ≥60 ml/min/1.73 m² with a need for additional glycemic control, the dose may be increased to 300 mg qd.
  In this study's dose-escalation phase, two dose levels will be evaluated:
  Low-dose cohort: 100 mg qd, taken before the first meal of the day. High-dose cohort: Starting dose of 100 mg qd for 1 week. If tolerated, the dose will escalate to 300 mg qd, taken before the first meal of the day.
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Low-dose cohort: 100 mg qd, taken before the first meal of the day. High-dose cohort: Starting dose of 100 mg qd for 1 week. If tolerated, the dose will escalate to 300 mg qd, taken before the first meal of the day.
  Other Names: ICIs

SUMMARY:
Colorectal cancer (CRC), ranking third in incidence among men and second in women globally with third-highest mortality in the US, remains a major health challenge despite multimodal therapies, particularly for advanced-stage patients with poor prognosis where immune checkpoint inhibitors (ICIs) like PD-1/PD-L1 blockers have emerged as transformative agents by reinvigorating anti-tumor immunity through PD-1/PD-L1 pathway inhibition. While MSI-H CRC's high mutational burden renders it susceptible to immunotherapy, clinical trials demonstrate durable responses with domestic ICIs such as tislelizumab showing 41.2% ORR, 14.4-month PFS, and 28.7-month OS in metastatic MSI-H CRC, yet unmet needs persist. Intriguingly, SGLT-2 inhibitor exhibit promising oncolytic potential, particularly when combined with ICIs, as evidenced by observational studies revealing enhanced tumor control in pancreatic ductal adenocarcinoma through metabolic-immunologic crosstalk and our preclinical data showing synergistic CRC growth suppression with the SGLT-2 inhibitor canagliflozin plus PD-1 blockade. This phase II trial investigates the safety and efficacy of canagliflozin-tislelizumab combination in metastatic MSI-H CRC, evaluating its impact on PFS, OS, and ORR while dissecting tumor microenvironment modulation mechanisms, thereby pioneering a novel metabolic-immunotherapy paradigm that could redefine treatment paradigms through dual metabolic-immune regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤80 years old at the time of signing the written informed consent form, regardless of gender.
2. Patients with histologically or cytologically confirmed colorectal cancer, including:

   1. Patients with unresectable locally advanced, recurrent, or distant metastatic colorectal cancer.
   2. Patients with wild-type RAS/RAF and BRAF V600E genotypes in tumor tissues.
   3. Patients with microsatellite instability-high (MSI-H) colorectal cancer confirmed by MSI testing.
   4. Patients who have experienced disease progression after receiving at least two lines of standard treatment, or who cannot tolerate the toxic side effects.
3. According to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), patients must have at least one target lesion with measurable diameters (tumor lesions with a long diameter ≥10 mm on CT scan, lymph node lesions with a short diameter ≥10 mm on CT scan, and a scan slice thickness of no more than 5 mm). Lesions that have received local treatments such as radiotherapy can be used as target lesions after clear progression is confirmed.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1, with an expected survival period of ≥3 months.
5. Patients must be type 2 diabetes mellitus (T2DM) patients and meet the indications for canagliflozin; or patients have no diagnosis of diabetes, no history of type 1 diabetes or diabetic ketoacidosis.

   The diagnosis of type 2 diabetes mellitus is defined as typical diabetic symptoms plus random blood glucose ≥11.1 mmol/L, or plus fasting blood glucose ≥7.0 mmol/L, or plus 2-hour post-load blood glucose in oral glucose tolerance test (OGTT) ≥11.1 mmol/L, or plus HbA1c ≥6.5%. For those without typical diabetic symptoms, reexamination on another day is required for confirmation (excluding random blood glucose).
6. Good function of major organs, that is, the relevant examination indicators within 14 days before randomization meet the following requirements (without blood or blood product transfusion, without the use of hematopoietic stimulating factors, and without the use of albumin or blood products):

   * Routine blood test: Hemoglobin ≥80 g/L; neutrophil count >1.5×10⁹/L; platelet count ≥90×10⁹/L.
   * Biochemical test: Total bilirubin ≤1.5×ULN (upper limit of normal value); serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN; serum creatinine (SCr) ≤1.5×ULN or creatinine clearance rate ≥50 mL/min (Cockcroft-Gault formula).
   * Prothrombin time (PT), international normalized ratio (INR) ≤1.5×ULN (unless warfarin anticoagulation is being used).
   * Cardiac Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥50%.
   * Renal function: eGFR ≥60 mL/min/1.73 m².
   * Blood glucose: HbA1c ≤9%.
7. Patients of childbearing potential (both male and female) must use effective medical contraceptive measures during the study period and within 6 months after the end of drug administration.
8. Body mass index (BMI) ≥18.5 kg/m² during the study screening period.
9. If complicated with hypertension, blood pressure must be controlled to a stable level with other medications.
10. No history of peripheral vascular disease, neuropathy, or diabetic foot ulcers.
11. Patients voluntarily join this study, sign the informed consent form, have good compliance, and patients and their families agree to cooperate with survival follow-up.

Exclusion Criteria:

1. Participation in other drug clinical trials within 4 weeks.
2. History of other tumors, except for in-situ cervical cancer, treated cutaneous squamous cell carcinoma, bladder epithelial tumors, or other malignant tumors that have received radical treatment (at least 5 years prior to enrollment).
3. Patients with symptomatic or rapidly progressive central nervous system metastases, extensive lung metastases causing dyspnea, or tumors approaching or invading major blood vessels or nerves.
4. Uncontrolled cardiac clinical symptoms or diseases, such as heart failure of NYHA class 2 or above, unstable angina, myocardial infarction within 1 year, or clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
5. Pregnant or lactating women.
6. Patients with active tuberculosis, bacterial or fungal infections (≥ grade 2, based on NCI-CTCAE 5.0), or HIV infection.
7. Patients with a history of psychoactive drug abuse that cannot be 戒除 (abstained from) or with mental disorders.
8. Subjects with any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: uveitis, enteritis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or childhood asthma that has fully remitted and requires no intervention in adulthood may be included; subjects with asthma requiring medical intervention with bronchodilators shall not be included).
9. Previous treatment with SGLT2 inhibitors (such as dapagliflozin, empagliflozin, canagliflozin).
10. Long-term steroid use or combined use of insulin/insulin sensitizers.
11. Baseline HbA1c >10%, history of stroke or transient ischemic attack within 5 years, and uncontrolled comorbidities.
12. Female subjects with a pregnancy plan or male subjects whose partners have a pregnancy plan from the screening period to 12 months after medication.
13. CRC patients with known BRAF V600E mutation or peritoneal cancer patients.
14. Patients with type 1 diabetes or diabetic ketoacidosis.
15. History of peripheral vascular disease, neuropathy, or diabetic foot ulcers.
16. Patients with severe renal insufficiency (eGFR <30 mL/min/1.73 m²).
17. Patients with recurrent genitourinary infections within six months or requiring long-term anti-infective treatment.
18. Patients with a history of lower limb amputation, severe peripheral vascular disease, or neuropathy.
19. Patients with uncontrolled hypothyroidism.
20. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Effect | through study completion, an average of 1 year
  Adverse Effect

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol